CLINICAL TRIAL: NCT07046468
Title: Measurement of Oxidation Reduction Potential in the Colon Using an Ingestible Sensor in Patietns With Ulcerative Colitis (UC) and Colorectal Cancer (CRC)
Brief Title: Smart Pill for Measuring Gut Health in Colon Inflammation and Colon Cancer
Acronym: SPIRIT
Status: Recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Stichting IMEC-NL (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-17771; NL88151.091.24 (Other: Netherlands Trial Register (NTR))
Record Dates: First submitted 2025-03-26; First posted 2025-07-01 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-02

CONDITIONS: Ulcerative Colitis (UC); Colorectal Cancer (CRC)
Keywords: Ulcerative Colitis; Colorectal cancer; Sensor; Redox; Oxidation reduction potential; Ingestible; Sensor pill; Inflammatory bowel disease
MeSH Terms: conditions — Colitis, Ulcerative; Colorectal Neoplasms; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ulcerative colitis
  Interventions: Device: Ingestion of sensor capsule (twice); Behavioral: Device evaluation questionnaire; Device: Wearing device; Behavioral: Monitoring sensor capsule exit; Device: Placement of devices at home; Diagnostic Test: Follow-up intestinal ultrasound
- Colorectal cancer
  Interventions: Device: Ingestion of sensor capsule (twice); Behavioral: Device evaluation questionnaire; Device: Wearing device; Behavioral: Monitoring sensor capsule exit; Device: Placement of devices at home

INTERVENTIONS:
Device: Ingestion of sensor capsule (twice) — Ingestion of the GISMO GEN1 System, an ingestible sensor capsule which measures pH, temperature and oxidation reduction potential (ORP) in the intestines.
  Other Names: GISMO GEN1 System
Behavioral: Device evaluation questionnaire — A 16-item online questionnaire to assess participant's experiences with the ingestible sensor capsule after the study measurements.
Device: Wearing device — Participants will wear a small device on a soft belt around their waist during study measurements with the sensor capsules.
Behavioral: Monitoring sensor capsule exit — Participants are instructed to press a button on the wearable device when they use the toilet for defaecation and wait with flushing to toilet until the wearable device indicates (using colored LEDs) that the toilet can be flushed and 1) that the sensor capsule is still in the body and study measurements continue or 2) that the sensor capsule has likely been excreted via the feces and the participant has to contact the research team to confirm exit.
Device: Placement of devices at home — Participants do not have to wear the device around the waist during sleeping. For optimal monitoring of sensor capsule exit during the nights, a second device will be placed on the participant's bedside table/close to the bed and a third device will be placed close to the toilet that the participant usually uses during the night.
Diagnostic Test: Follow-up intestinal ultrasound — At 3 months after treatment initiation, participants with ulcerative colitis will undergo a follow-up intestinal ultrasound (IUS) (non-endoscopic) outside of routine care to assess treatment response.
  Groups: Ulcerative colitis

SUMMARY:
The goal of this observational pilot study with invasive measurements is to explore whether an ingestible sensor pill can be of use in diagnosis or monitoring of disease in patients with ulcerative colitis or colorectal cancer. The main questions it aims to answer are:

* which changes in bowel environment can the sensor pill measure in ulcerative colitis and colorectal cancer before and after treatment?
* how practical, effective and user-friendly is the sensor pill for measuring bowel environment in patients with bowel disease?

Participants will:

* take one sensor pill before treatment and take one sensor pill three months after (start of) treatment;
* monitor sensor pill bowel exit using a small wearable device;
* answer a questionnaire on experience with the sensor pill;
* receive an extra bowel ultrasound (non-endoscopic) three months after start of treatment (only for participants with ulcerative colitis).

DETAILED DESCRIPTION:
Rationale: The gold standard diagnostic tool for inflammatory bowel disease (IBD) and colorectal carcinoma (CRC) is endoscopy, which can be burdensome for patients. The future of IBD care demands novel, minimally invasive biomarkers for personalized care and CRC screening programs could greatly benefit from new minimally invasive diagnostic tools. Oxidative stress plays a significant role in the progression of gut inflammation and colorectal cancer. Using an ingestible sensor, we aim to measure oxidation-reduction potential (ORP) directly in the gut. We hypothesize that it is feasible to measure intestinal ORP with an ingestible sensor and expect that ORP levels are elevated in patients with active ulcerative colitis (UC) and CRC before treatment, compared to after treatment.

Objective: Measurement of intestinal oxidation-reduction potential using a smart sensing ingestible and its relation to active UC and CRC.

Study design: Observational, exploratory study with invasive measurements.

Study population: 5 patients ≥ 18 years of age with UC and 5 patients ≥ 18 years of age with CRC

Main study parameters/endpoints: The main study parameter is colonic ORP profiles measured with the ingestible sensor ingestible compared before and after treatment for UC and CRC.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Risk associated with participation are deemed low. Medical or surgical treatment is not altered in any way. Patients with UC will receive an additional IUS. The GISMO GEN1 ingestible device (size 21.8 mm x 7.64 mm) is an investigational tool deemed safe for human use in clinical settings, with risks detailed in the IMDD. Device exit will be tracked via the temperature sensor of the ingestible sensor. If exit is not confirmed after 14 days, an X-ray will confirm whether the device is still in the gastrointestinal tract. If visible on the X-ray, a medical specialist will determine further action, which may include laxatives or surgery, with costs covered by the research team. If X-ray examination is necessary, the participant may experience a maximum radiation exposure of 0.10 mSv. Participant burden is low; time investment including study visits, device checks and questionnaire is estimated around 4 hours in total. Main burden is expected to be the continuous wearing of the base device as long as the ingestible sensor remains in the body.

ELIGIBILITY:
Inclusion Criteria:

(For all participants:)

* Age ≥ 18 years old;
* willing and able to provide informed consent;
* defaecation pattern: generally at least one defaecation per 48 hours.

(For the UC group:)

* Diagnosis of UC confirmed by clinical, endoscopic, and/or histological evidence prior to screening as per standard criteria;
* moderately to severely active UC determined by intestinal ultrasound (bowel wall thickness (BWT) > 3 mm), starting treatment or requiring change in treatment due to non-response to their existing treatment;
* starting or optimizing treatment for colitis (including aminosalicylates, oral corticosteroids, thiopurines, biologics and small molecules).

(For the CRC group:)

* Diagnosis of non-obstructing non-locally advanced colorectal adenocarcinoma;
* ready/planned for surgery of CRC.

Exclusion Criteria:

(For all participants:)

* Body mass index (BMI) > 30 kg/m^2;
* known obstruction, stricture or stenosis in the gastrointestinal tract not attributable to current inflammation or tumour, potentially blocking ingestible passage. Determined as per discretion of gastroenterologist/oncologist using standard procedural clinical diagnostic or imaging techniques;
* history of complex bowel resection or recent intra-abdominal surgery (< 3 months);
* known abdominal adhesions;
* swallowing disorders, including achalasia or oropharyngeal dysfunction;
* ongoing infections;
* known to be pregnant, lactating or actively trying to get pregnant (self-reported);
* short bowel syndrome or ostomy;
* only parenteral diet;
* pacemaker or other implantable electronic devices;
* planned magnetic resonance imaging (MRI) procedure during the ingestible meaurement period;
* unwilling to undergo an X-ray examination (in the case ingestible exit cannot be confirmed);
* participation in other medical interventional/Wet medisch-wetenschappelijk onderzoek (WMO)-compliant reearch;
* participant is working (as medical personnel) in a professional healthcare facility (intensive care, emergency room, surgery rooms, clinics, patient rooms), military area (e.g. submarine, near radar installation), or heavy industrial area (e.g. power plants, automotive, mining, refineries) during the duration of the clinical investigation.

(For the CRC group:)

* Diagnosis or strong suspicion of IBD;
* planned treatment with adjuvant chemotherapy or radiotherapy.

(For the UC population:)

* Diagnosis or strong suspicion of colorectal adenocarcinoma;
* use of rectal foam/enema during the measurement period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be performed in outpatients ≥18 years old. Five patients will be included with moderately to severely active UC, starting new treatment; five patients with colorectal adenocarcinoma, planned for surgery.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Intestinal ORP measurements | Baseline and at 3 months after start of treatment.
  ORP profile in the colon using the GISMO GEN1 System in patients with UC or CRC.
Disease activity (SCCAI) | Baseline and 3 months after start of treatment.
  UC disease activity as determined by the Simple Clinical Colitis Activity Index
Disease activity (FC) | Baseline and at 3 months after treatment start.
  UC disease activity as determined by the faecal calprotectin (in microgram/gram)
Tumor stage | Directly after surgical resection
  TNM tumor stage as recorded in pathology report.
Tumor size | Directly after surgical resection
  Tumor size as recorded in surgery report.
Tumor resection margin status | Directly after surgical resection
  Residual tumor at the primary site after surgical resection as classified in pathology report.
Tumor differentiation grade | Directly after surgical resection
  Tumor differentiation grade as recorded in pathology report.

SECONDARY OUTCOMES:
Intestinal pH | From enrollment to 3 months after start of treatment.
  Intestinal pH measured with the ingestible sensor capsule.
Area of inflammation | Directly after intestinal ultrasound.
  Area of inflammation in patients with UC, as recorded in the intestinal ultrasound report.
Tumour location | Directly post-surgery.
  Tumor location in patients with CRC as recorded in the surgery report.
Ingestible transit time. | Baseline and at 3 months after start of treatment.
  Time from ingestion to defaecation in hours.
Data coverage | Baseline and at 3 months after start of treatment
  Data coverage of recordings with the ingestible sensor capsule in minutes of data recorded as percentage of transit time in minutes (%)
Participant experience | Up to 1 month after exit of the post-treatment ingestible sensor capsule measurement period.
  Participant experience determined with a satisfaction questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Marjolijn Duijvestein, MD PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No
The data that supports the findings of this study can be made available upon request to the corresponding author within the regulations of the applicable regulations and ethical considerations.